CLINICAL TRIAL: NCT02312180
Title: A Phase 1, Dose Escalation, and Pharmacokinetic Study of ProMetic Plasminogen Administered as Intravenous Infusion in Adults and Children With Hypoplasminogenemia
Brief Title: A Phase 1 Study of ProMetic Plasminogen (Human) Intravenous in Adults and Children With Plasminogen Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prometic Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002C005G
Expanded Access: NCT03265171 (No longer available)
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Type I Plasminogen Deficiency; Hypoplasminogenemia
MeSH Terms: conditions — Plasminogen Deficiency, Type I; Congenital Plasminogen Deficiency | interventions — Plasminogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): low dose group of 2 mg/kg Plasminogen (Human) Intravenous
  Interventions: Biological: Plasminogen (Human) Intravenous
- Cohort 2 (Experimental): mid-dose group of 6 mg/kg Plasminogen (Human) Intravenous
  Interventions: Biological: Plasminogen (Human) Intravenous

INTERVENTIONS:
Biological: Plasminogen (Human) Intravenous — Plasma-derived purified plasminogen formulated for intravenous administration

SUMMARY:
ProMetic is intiitating a first-in-man study entitled "A Phase 1, Dose Escalation, and Pharmacokinetic Study of ProMetic Plasminogen Administered as Intravenous Infusion in Adults and Children with Hypoplasminogenemia". The general objectives of this clinical study, (Protocol #2002C005G), are to determine the optimal dose and interval required to support the planned Phase 2/3 study and to investigate initial safety and tolerability.

DETAILED DESCRIPTION:
The Phase 1 study will be a single center study, the subjects will be from across country. It is an open-label, single-arm, dose-escalation study in patients with hypoplasminogenemia aged 12 years and older.

Three dose cohorts are planned to achieve a target sample size of 12 evaluable subjects. This will ensure a minimum of 4 evaluable subjects in each cohort. Due to the challenges of patient availability and burden of cross country travel, each cohort will enroll no more than 6 subjects. Any subject may participate in multiple cohorts, as judged appropriate by the investigator.

In each cohort, each subject must be diagnosed with hypoplasminogenimia and have a plasminogen activity level of ≤ 40% before they will be administered a single dose of Plasminogen (Human), the investigational medicinal product. Plasminogen will be administered as an intravenous (IV) infusion at the following doses:

* Cohort 1: 2 mg/kg
* Cohort 2: 6 mg/kg
* Cohort 3*: 12 mg/kg * Optional. If optimal dosing information is demonstrated in either Cohort 1 or 2, Cohort 3 will not be pursued.

At each dose level, Plasma plasminogen activity and antigen levels will be measured to develop a pharmacokinetic profile. Blood samples will be drawn at the following time points: baseline immediately before dosing; at the end of infusion; and at 1, 6, 24, 48, 72, 96, 120, 168, and 216 hours after the end of infusion. Visits 1-4 and 11 must be conducted at the clinical site. A subject may conduct Visits 5-10 at the clinical site or have the study procedures performed by a Home Health Nurses Group (HHNG) nurse through home visits, if continued visits to the study site are not possible or practical.

Subjects will have another visit 14 days after the IV infusion for Visit 10 (Day 15, Short-term-Safety Visit). Subjects will return to the clinic 30 days after IV infusion for Visit 11 (Day 30, Follow-up-Safety Visit) for the collection of adverse events (AEs), immunogenicity testing, routine safety tests and procedures, and final viral safety testing, unless the subject is entering into another Cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided informed consent/assent, or the subject's guardian has given consent if the subject is under 18 years
2. Subject is male or female between 12 and 80 years of age, inclusive
3. Subject has a diagnosis of hypoplasminogenemia evidenced by an abnormal, decreased plasminogen activity level, regardless of plasminogen antigen level
4. Subject has a plasminogen activity level ≤ 40%
5. Subject has documented immunity to hepatitis A virus (HAV) and hepatitis B virus (HBV) or has received the first dose of HAV and HBV vaccine prior to IMP administration and is scheduled to receive the second vaccine dose
6. Subject (male or female of reproductive age) agrees to use contraceptive methods from screening through 14 days after administration of IMP unless documented as biologically (e.g., post-menopausal, not begun menstruating) or surgically (vasectomized) sterile

Exclusion Criteria:

1. Subject has a history of severe reactions (e.g., anaphylaxis) to blood or blood products that may requiring resuscitation or otherwise prevent study participation in the opinion of the investigator
2. Subject has evidence of uncontrolled hypertension
3. Subject has clinical or laboratory evidence of an intercurrent infection as evidenced by symptoms including fever, tachycardia, or other specific signs and symptoms*
4. Subject is pregnant and/or lactating
5. Subject has or has had a malignancy, except for basal and squamous cell skin cancer, within 3 years of Baseline
6. Subject is a previous organ transplant recipient
7. Subject is receiving exogenous plasminogen (ocular or IV), including laboratory grade plasminogen and fresh lyophilized plasma within two weeks of Baseline
8. Subject has any psychiatric disorder, other mental disorder, or any other medical disorder that impairs the subject's ability to give informed consent or to comply with the requirements of the study protocol
9. Subject has experienced a severe adverse event in a prior cohort of this study.
10. Subject has evidence of renal dysfunction, defined as serum creatinine of > 2 times the upper limit of normal
11. Subject has evidence of hepatic dysfunction, defined as 3 times the upper limit of normal in ALT, and/or AST, and/or alkaline phosphatase (ALP)
12. Subject has participated in another IRB-approved interventional clinical trial of a drug, biologic, or device within 30 days of Baseline
13. Subject has a chronic or acute, clinically significant, inter-current illness (eg, cardiac, hepatic, renal, endocrine, neurologic, hematologic, neoplastic, immunological, and skeletal) that the investigator determines could interfere with the safety or pharmacokinetic assessments for this study
14. Subject is unable to adhere to the scheduling requirements of the protocol *Note: Subjects with an intercurrent infection cannot participate; however, subjects meeting this exclusion criterion at the Baseline Visit may return for a repeat Baseline Visit once the infection is considered resolved according to the investigator and can be included in the cohort that is actively recruiting at that time if all inclusion/exclusion criteria are met

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profile of lyophilized plasminogen (PLG). Area under the concentration time curve (both AUC0-t and AUC0-inf), maximum plasma concentration (Cmax), volume of distribution (Vd), clearance (Cl), and mean residence time (MRT). | 8 months
  The following PK parameters will be calculated from PLG activity and antigen levels using the non-compartmental PK analysis method: Area under the concentration time curve (both AUC0-t and AUC0-inf), maximum plasma concentration (Cmax), volume of distribution (Vd), clearance (Cl), and mean residence time (MRT). Pharmacokinetic (PK) profile of lyophilized plasminogen (PLG) at 3 dose levels (the third dose is optional) in subjects with hypoplasminogenemia to determine the desirable dose and dosing interval to be studied in a Phase 2/3 study.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of PLG in subjects with hypoplasminogenemia, as measured by Rate, severity, and relatedness of any adverse events. | 8 months
  Rate, severity, and relatedness of any adverse events. Changes from baseline observed or reported in medical history, vital signs, physical exam, clinical laboratory tests. Assessment of development of antibodies against plasminogen.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana Hemophilia and Thrombosis Center, Indianapolis, Indiana, United States